CLINICAL TRIAL: NCT02194101
Title: Supernormal Oxygen Delivery May Not be a Valid Goal for Patients With Proximal Femur Fracture. An Observational Pilot Study
Brief Title: Supernormal Goal for Proximal Femur Fracture
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Xiangcai Ruan, Vice-Chair, Guangzhou First People's Hospital
Other Study IDs: GZFPH-IRB-2013-049
Record Dates: First submitted 2014-07-14; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Femoral Fractures
Keywords: oxygen delivery; proximal femoral fracture; goal-directed therapy
MeSH Terms: conditions — Femoral Fractures; Proximal Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Supernormal oxygen delivery goal therapy: Patients will be aged over 70 yr and weight over 35 kg, and undergoing proximal femur fracture (PFF) surgery under peripheral nerve block and laryngeal mask airway anesthesia.
  Interventions: Procedure: Supernormal oxygen delivery goal therapy

INTERVENTIONS:
Procedure: Supernormal oxygen delivery goal therapy — A 10% increase in stroke volume (SV) after fluid challenge (5 ml/kg) with Ringer's lactate solution will be deemed positive. Oxygen delivery will be check when fluid challenge becomes negative. If oxygen delivery index (DO2I) can not be greater than 600 mL/m2, then dobutamine will be started at a dose of 2.5 μg/kg/min and increased by the same increment every 20 minutes until the described target is reached or until a maximal dose of 10 μg/kg/min is given. Dobutamine is decreased in dose or discontinued if the heart rate is above 100 beats per minute or shows signs of cardiac ischemia. Blood transfusions will be used to maintain a hemoglobin concentration over 8mg/dL.

SUMMARY:
This is an observational pilot study of supernormal oxygen delivery goal for patients with proximal femoral fracture.

DETAILED DESCRIPTION:
Augmentation of oxygen delivery using fluids with or without inotropes has been shown to improve surgical outcome in high-risk patients. Patients with proximal femoral fracture are considered high risk. However, most of this cohort elderly patients have poor cardiovascular condition and may not achieve the oxygen delivery goal. We will perform an observational pilot study whether the supernormal oxygen delivery is a valid hemodynamic goal for patients with proximal femoral fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 70 yr
* Weight over 35 kg
* Underwent proximal femur fracture (PFF) surgery under peripheral nerve block and laryngeal mask airway anesthesia.

Exclusion Criteria:

* Patients who could be harmed due to the treatment (ongoing myocardial infarction, chronic dialysis)
* Monoamine oxidase inhibitor use within the last 14 days
* Pathological fractures and conditions
* Inability to give informed consent(as judged by a research team member)
* Anticipated difficulties obtaining data during the first postoperative year (as judged by a research team member)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients will be aged over 70 yr and weight over 35 kg, and undergoing proximal femur fracture (PFF) surgery under peripheral nerve block and laryngeal mask airway anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Oxgen delivery index | At the end of 4 hour goal-directed therapy
  To attain a improved oxygen delivery index at the end of 4 hour goal-directed therapy

SECONDARY OUTCOMES:
Hear rate augmentation | Day 1
Hemodynamic response | Day 1
  Including stroke volume, cardiac index, base excess, lactate, hemoglobin, and urine output.
fluid volume administrated | intraoperatively
Length of hospital stay | Day 30
Postoperative morbidity | day 5

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcai Ruan, MD., PhD., Principal Investigator — Guangzhou First Municipal People's Hospital,Guangzhou,Guangdong,China,510180
Locations (1):
- Guangzhou First Municipal People's Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Pestana D, Espinosa E, Eden A, Najera D, Collar L, Aldecoa C, Higuera E, Escribano S, Bystritski D, Pascual J, Fernandez-Garijo P, de Prada B, Muriel A, Pizov R. Perioperative goal-directed hemodynamic optimization using noninvasive cardiac output monitoring in major abdominal surgery: a prospective, randomized, multicenter, pragmatic trial: POEMAS Study (PeriOperative goal-directed thErapy in Major Abdominal Surgery). Anesth Analg. 2014 Sep;119(3):579-587. doi: 10.1213/ANE.0000000000000295. PMID 25010820
- [Result] Bennett-Guerrero E. Hemodynamic goal-directed therapy in high-risk surgical patients. JAMA. 2014 Jun 4;311(21):2177-8. doi: 10.1001/jama.2014.5306. No abstract available. PMID 24841970
- [Result] Salzwedel C, Puig J, Carstens A, Bein B, Molnar Z, Kiss K, Hussain A, Belda J, Kirov MY, Sakka SG, Reuter DA. Perioperative goal-directed hemodynamic therapy based on radial arterial pulse pressure variation and continuous cardiac index trending reduces postoperative complications after major abdominal surgery: a multi-center, prospective, randomized study. Crit Care. 2013 Sep 8;17(5):R191. doi: 10.1186/cc12885. PMID 24010849
- [Result] Bartha E, Arfwedson C, Imnell A, Fernlund ME, Andersson LE, Kalman S. Randomized controlled trial of goal-directed haemodynamic treatment in patients with proximal femoral fracture. Br J Anaesth. 2013 Apr;110(4):545-53. doi: 10.1093/bja/aes468. Epub 2012 Dec 28. PMID 23274782
- [Result] Cecconi M, Fasano N, Langiano N, Divella M, Costa MG, Rhodes A, Della Rocca G. Goal-directed haemodynamic therapy during elective total hip arthroplasty under regional anaesthesia. Crit Care. 2011;15(3):R132. doi: 10.1186/cc10246. Epub 2011 May 30. PMID 21624138
- [Result] Davies SJ, Yates D, Wilson RJ. Dopexamine has no additional benefit in high-risk patients receiving goal-directed fluid therapy undergoing major abdominal surgery. Anesth Analg. 2011 Jan;112(1):130-8. doi: 10.1213/ANE.0b013e3181fcea71. Epub 2010 Nov 3. PMID 21048092
- [Result] Grocott MP, Dushianthan A, Hamilton MA, Mythen MG, Harrison D, Rowan K; Optimisation Systematic Review Steering Group. Perioperative increase in global blood flow to explicit defined goals and outcomes after surgery: a Cochrane Systematic Review. Br J Anaesth. 2013 Oct;111(4):535-48. doi: 10.1093/bja/aet155. Epub 2013 May 9. PMID 23661403
- [Result] Bisgaard J, Gilsaa T, Ronholm E, Toft P. Optimising stroke volume and oxygen delivery in abdominal aortic surgery: a randomised controlled trial. Acta Anaesthesiol Scand. 2013 Feb;57(2):178-88. doi: 10.1111/j.1399-6576.2012.02756.x. Epub 2012 Aug 17. PMID 22897633